CLINICAL TRIAL: NCT06851533
Title: Comparison of the Effects of Thoracolumbar Interfascial Plane Block and Quadro Iliac Plane Block on Postoperative Opioid Consumption After Lumbar Microsurgery: A Randomized Controlled Trial
Brief Title: Comparing Thoracolumbar Interfascial and Quadro Iliac Plane Blocks on Postoperative Opioid Use Following Lumbar Microsurgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Burak Omur, Assistant Professor, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lumbar tlip vs quadroilaac
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Microdiscectomy; Nerve Block
Keywords: Postoperative pain; Ultrasound-guided nerve block
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Block (Control Group) (Active Comparator): Patients receive standard perioperative analgesia without any additional regional block.
  Interventions: Procedure: Standard Analgesia (No Block)
- TLIP Block (Experimental): Patients receive the Thoracolumbar Interfascial Plane (TLIP) block in addition to standard perioperative analgesia.
  Interventions: Procedure: Thoracolumbar Interfascial Plane (TLIP) Block
- Quadro Iliac Plane Block (Experimental): Patients receive the Quadro Iliac Plane Block in addition to standard perioperative analgesia.
  Interventions: Procedure: Quadro Iliac Plane Block

INTERVENTIONS:
Procedure: Standard Analgesia (No Block) — Participants receive standard perioperative analgesia (including intravenous paracetamol/tramadol), but no additional regional block is applied.
  Arms: No Block (Control Group)
Procedure: Thoracolumbar Interfascial Plane (TLIP) Block — In addition to standard perioperative analgesia, a TLIP block is performed under sterile conditions and ultrasound guidance, after the surgical procedure is completed but before the patient is awakened. A total of 20 mL of 0.25% bupivacaine is injected into the thoracolumbar fascial plane, and spread is confirmed via ultrasound.
  Arms: TLIP Block
Procedure: Quadro Iliac Plane Block — In addition to standard perioperative analgesia, a Quadro Iliac Plane Block is performed under sterile conditions and ultrasound guidance, after the surgical procedure is completed but before the patient is awakened. A total of 20 mL of 0.25% bupivacaine is injected into the quadro iliac plane at the level of the iliac crest, and spread is confirmed via ultrasound.
  Arms: Quadro Iliac Plane Block

SUMMARY:
Lumbar microdiscectomy is a commonly used surgical procedure for treating herniated discs. Effective postoperative analgesia is crucial for early mobilization and functional recovery. Uncontrolled postoperative pain can delay recovery, increase the risk of opioid dependence, and lead to respiratory complications.

Although opioid analgesics effectively reduce pain, they can cause side effects such as nausea, vomiting, respiratory depression, and dependency. Therefore, non-opioid analgesic methods are preferred for patient safety and comfort. Recently, regional anesthesia techniques such as the Thoracolumbar Interfascial Plane (TLIP) block and the Quadro Iliac Plane Block have been introduced for postoperative pain management in lumbar surgeries. However, there are not enough studies comparing the superiority of these two methods.

Study Objective: The primary aim of this study is to evaluate the effects of ultrasound-guided TLIP and Quadro Iliac Plane Blocks on postoperative opioid consumption after lumbar microsurgery. The secondary aim is to compare opioid-related side effects (such as nausea, vomiting, respiratory depression, etc.) and postoperative NRS pain scores between the groups.

DETAILED DESCRIPTION:
Lumbar microdiscectomy is a widely performed surgical procedure for the treatment of lumbar disc herniation. Ensuring optimal analgesia during the postoperative period is crucial for promoting functional recovery and early mobilization. Inadequate control of postoperative pain may delay the healing process, increase the risk of opioid dependence, and lead to respiratory complications.

Although opioid analgesics are effective in alleviating pain during the postoperative period, they can cause adverse effects such as nausea, vomiting, respiratory depression, and an increased risk of dependence. Therefore, the implementation of non-opioid analgesic strategies is essential for maintaining patient safety and comfort. In recent years, regional anesthesia techniques, including the Thoracolumbar Interfascial Plane block and the Quadro Iliac Plane Block, have been utilized for postoperative pain management in lumbar surgeries. However, there is insufficient evidence directly comparing the effectiveness of these two methods.

Purpose of the Study: The primary objective of this study is to evaluate the impact of ultrasound-guided Thoracolumbar Interfascial Plane and Quadro Iliac Plane Blocks on postoperative opioid consumption following lumbar microsurgery. Additionally, the secondary objective is to compare the incidence of opioid-related side effects (such as nausea, vomiting, and respiratory depression) and patients' postoperative pain scores, measured using the Numeric Rating Scale, between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years
* American Society of Anesthesiologists (ASA) physical status I to III
* scheduled for lumbar microdiscectomy surgery

Exclusion Criteria:

* Known allergy to local anesthetics
* Any other significant drug allergies related to the study interventions
* Pregnancy
* Pre-existing psychiatric or neurological disorders
* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
tramadol consumption | first 24 hours after the operation
  Total tramadol consumption (mg) in the first 24 hours after surgery.

SECONDARY OUTCOMES:
NRS (Numerical Rating Scale) pain scores | first 24 hours after the operation
  NRS (0-10) scores will be measured at 3, 6, 12, 18, and 24 hours during both rest and mobilization in the postoperative period.
opioid-related side effects (such as nausea, vomiting, respiratory depression) | first 24 hours after the operation
  The incidence of opioid-related side effects (e.g., nausea, vomiting, respiratory depression) will be recorded and compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication

REFERENCES:
- [Background] Canikli Adiguzel S, Akyurt D, Bahadir Altun H, Ultan Ozgen G, Akdeniz S, Bayraktar B, Tulgar S, Yigit Y. Posterior Quadratus Lumborum Block or Thoracolumbar Interfascial Plane Block and Postoperative Analgesia after Spinal Surgery: A Randomized Controlled Trial. J Clin Med. 2023 Nov 21;12(23):7217. doi: 10.3390/jcm12237217. PMID 38068268
- [Background] Hu Z, Han J, Jiao B, Jiang J, Sun Y, Lv Z, Wang J, Tian X, Wang H. Efficacy of Thoracolumbar Interfascial Plane Block for Postoperative Analgesia in Lumbar Spine Surgery: A Meta-analysis of Randomized Clinical Trials. Pain Physician. 2021 Nov;24(7):E1085-E1097. PMID 34704718
- [Background] Yildirim Uslu E. Effect of Quadratus Lumborum Block in Patients With Acute-Subacute Unilateral Lumbar Strain. Cureus. 2024 May 24;16(5):e61014. doi: 10.7759/cureus.61014. eCollection 2024 May. PMID 38915966